CLINICAL TRIAL: NCT04729127
Title: A Randomized Trial of Project ImPACT, an Evidence-based Intervention for Infants and Toddlers With Autism Spectrum Disorder
Brief Title: A Trial of Project ImPACT in Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Melanie Pellecchia, PhD, Principal investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 842506
Record Dates: First submitted 2021-01-22; First posted 2021-01-28 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (No Intervention): The families keep receiving their treatment as usual
- ImPACT at a dose of 1 hour/week (Active Comparator): ImPACT at a dose of 1 hour/week over 6 months
  Interventions: Behavioral: Project ImPACT
- ImPACT at 4 hours/week (Active Comparator): ImPACT at 4 hours/week over 6 months.
  Interventions: Behavioral: Project ImPACT

INTERVENTIONS:
Behavioral: Project ImPACT — Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
  Arms: ImPACT at 4 hours/week; ImPACT at a dose of 1 hour/week

SUMMARY:
Our pilot study will address a number of pressing questions, including: Can community clinicians successfully coach parents of children with ASD in evidence-based practice to achieve positive outcomes for their children and themselves? What dose is necessary to achieve change? And what is the cost effectiveness of implementing evidence-based interventions at different doses?

DETAILED DESCRIPTION:
The investigators will partner with 6 of Philadelphias 13 agencies serving young children with ASD. The investigators will enroll 3 clinicians per agency (18 total) and 3 families per clinician (54 total). Agencies will be randomized to the 3 arms. The investigators will measure clinician fidelity and parent fidelity through direct observation and selfreport. The investigators will measure child and parent outcomes at baseline and 6 months using measures common to similar trials. Resource use for the economic evaluation will occur quarterly and will take a societal approach. The investigators will partner with a community advisory board to apply the findings from this pilot trial to the development of a larger, system-wide subsequent trial that is feasible and ecologically valid for Philadelphias EI system. The results will provide rigorous information about whether evidence-based autism interventions for young children can be implemented successfully with the resources available in cities like Philadelphia, the role of hours of treatment in improving child outcomes, and the cost-benefit implications for families and community agencies. This project has the potential to dramatically improve the services families of young children with ASD in Philadelphia receive, and significantly improve their long-term outcomes. This preliminary trial would provide the EI system with the information needed to bring this type of intervention to scale across the entire system. It also would serve as the foundation for an application for federal funds to conduct a system-wide study of Project ImPACT as implemented in all Philadelphia agencies serving children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. child is <30 months of age (to receive 6 months of intervention)
2. a classification of autism or high autism risk as determined by the EI system;
3. receive early intervention services through the infant and toddler program; and
4. parent is willing to complete the parent measures that are part of this study.

Exclusion Criteria:

1) be over 30 months of age

Max Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Mental Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Parent/Children dyads were enrolled in the study and counted as 1 family. The total number includes the number of individual parents and children enrolled together as a dyad and individual early intervention providers that were enrolled.
Groups:
- Treatment as Usual: Children; Treatment as Usual: Caregivers: The families keep receiving their treatment as usual.
- Treatment as Usual: Early Interventionists: Early interventionists provide services and treatments as they usually would.
- ImPACT at a Dose of 1 Hour/Week: Children; ImPACT at a Dose of 1 Hour/Week: Caregivers: ImPACT at a dose of 1 hour/week over 6 months
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at a Dose of 1 Hour/Week: Early Interventionists: Early interventionists provider ImPACT at a dose of 1 hour/week over 6 months to at least 3 families on their caseload.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at 4 Hours/Week: Children: ImPACT at 4 hours/week over 6 months.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at 4 Hours/Week: Early Interventionists: Early interventionists provider ImPACT at a dose of 4 hours/week over 6 months to at least 3 families on their caseload.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at a Dose of 4 Hours/Week: Caregivers: ImPACT at a dose of 4 hours/week over 6 months
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
Period: Overall Study
Arm/Group | Treatment as Usual: Children | Treatment as Usual: Early Interventionists | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Children | ImPACT at a Dose of 1 Hour/Week: Early Interventionists | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Children | ImPACT at 4 Hours/Week: Early Interventionists | ImPACT at a Dose of 4 Hours/Week: Caregivers
Started | 18 | 6 | 18 | 23 | 6 | 23 | 20 | 6 | 20
Completed | 12 | 6 | 12 | 16 | 6 | 16 | 17 | 6 | 17
Not Completed | 6 | 0 | 6 | 7 | 0 | 7 | 3 | 0 | 3
Not completed — Suspended/Terminated EI Services | 4 | 0 | 4 | 6 | 0 | 6 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Switched Agency/Setting | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Sex/gender was not collected for caregiver participants in all treatment groups. The sociodemographic form did not contain questions about the sex/gender of caregiver participants, and their overall count for this section will be 0.
Groups:
- Treatment as Usual: Early Interventionists: Early interventionists provide treatment and services as usual.
- ImPACT at a Dose of 1 Hour/Week: Early Interventionists: Early Interventionists provide ImPACT at a dose of 1 hour/week over 6 months with at least 3 families on their caseload.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at 4 Hours/Week: Early Interventionists: Early Interventionists provide ImPACT at a dose of 4 hours/week over 6 months with at least 3 families on their caseload.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at 4 Hours/Week: Caregivers: ImPACT at 4 hours/week over 6 months.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual: Children | Treatment as Usual: Early Interventionists | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Children | ImPACT at a Dose of 1 Hour/Week: Early Interventionists | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Children | ImPACT at 4 Hours/Week: Early Interventionists | ImPACT at 4 Hours/Week: Caregivers | Total
Number analyzed (Participants) | 18 | 6 | 18 | 23 | 6 | 23 | 20 | 6 | 20 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 0 | 0 | 23 | 0 | 0 | 20 | 0 | 0 | 61
  Between 18 and 65 years | 0 | 6 | 18 | 0 | 6 | 23 | 0 | 6 | 20 | 79
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.92 (0.42) | 42.4 (9.66) | 28.9 (5.9) | 1.86 (0.48) | 42.2 (9.24) | 32.0 (7.2) | 2.02 (0.26) | 39.5 (8.71) | 35.8 (9.6) | 10.74 (16.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Data on sex/gender was collected through a sociodemographic survey. The sociodemographic survey did not ask for sex/gender information for caregivers across the three arms. Results are only available for children and early interventionists. Population: Sex/gender was not collected for caregiver participants in all treatment groups. The sociodemographic form did not contain questions about the sex/gender of caregiver participants. The overall count will be 0 for caregiver participants across treatment groups.
  Participants
    number analyzed (Participants) | 18 | 6 | 0 | 23 | 6 | 0 | 20 | 6 | 0 | 79
    Female | 8 | 4 | 0 | 6 | 6 | 0 | 8 | 6 | 0 | 38
    Male | 10 | 2 | 0 | 17 | 0 | 0 | 12 | 0 | 0 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Asian | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 9 | 1 | 6 | 9 | 3 | 12 | 10 | 2 | 9 | 61
  White | 5 | 3 | 5 | 7 | 3 | 6 | 3 | 4 | 4 | 40
  More than one race | 0 | 0 | 3 | 2 | 0 | 4 | 1 | 0 | 1 | 11
  Unknown or Not Reported | 1 | 1 | 1 | 3 | 0 | 0 | 5 | 0 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 18 | 23 | 6 | 23 | 20 | 6 | 20 | 140

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales 3rd Edition-Communication Domain
Description: The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.
  Because it is a norm-based instrument, the examinee's adaptive functioning is compared to that of others his or her age. The ABC score is based on scores for three specific adaptive behavior domains: Communication, Daily Living Skills, and Socialization.
  The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The standard score range for the Communication domain is 20-140. Higher scores indicate better outcomes.
Time Frame: Time 1 (Baseline) and Time 3 (6 Month Follow Up) for a total of 6 months.
Population: Participants in the arms/groups "Treatment as Usual: Early Interventionists", "ImPACT at a Dose of 1 Hour/Week: Early Interventionists", "ImPACT at 4 Hours/Week: Early Interventionists", "Treatment as Usual: Caregivers", "ImPACT at a Dose of 1 Hour/Week: Caregivers", and ImPACT at 4 Hours/Week: Caregivers" are not included in the analysis as the measure's intent is to assess child outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | ImPACT at a Dose of 1 Hour/Week | ImPACT at 4 Hours/Week
Number analyzed (Participants) | 12 | 17 | 17
units on a scale
  Baseline | 69.4 (15.2) | 65.2 (14.0) | 63.4 (18.0)
  Follow-Up | 69.4 (15.7) | 61.4 (21.6) | 54.9 (18.4)
Statistical Analysis 1: Comparison: Treatment as Usual vs ImPACT at a Dose of 1 Hour/Week; See protocol for full statistical analysis plan; Test type: Other; p = .79, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual vs ImPACT at 4 Hours/Week; See protocol for full statistical analysis plan; Test type: Other; p = .27, Regression, Linear

2. Primary Outcome: Brief Observation of Social Communication Change (BOSCC)
Description: The BOSCC is a measure of treatment-response for social-communication behaviors.
  The BOSCC contains 12 items in total. The score range of individual items is 0-5. Items are then summed to a total score. The range for a total score is 0-60. Higher scores are an indication of more symptom severity.
Time Frame: Baseline and 6 Month Follow Up (Exit) (6 months)
Population: Participants in the arms/groups "Treatment as Usual: Early Interventionists", "ImPACT at a Dose of 1 Hour/Week: Early Interventionists", "ImPACT at 4 Hours/Week: Early Interventionists", "Treatment as Usual: Caregivers", "ImPACT at a Dose of 1 Hour/Week: Caregivers", "ImPACT at 4 Hours/Week: Caregivers" are not included in the analysis as the measure's intent is to assess child outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual: Children | ImPACT at a Dose of 1 Hour/Week: Children | ImPACT at 4 Hours/Week: Children
Number analyzed (Participants) | 12 | 17 | 17
score on a scale
  Baseline | 35.6 (29.2) | 36.6 (8.5) | 37.0 (8.8)
  Follow-Up | 29.2 (10.3) | 34.8 (10.3) | 36.2 (5.6)
Statistical Analysis 1: Comparison: Treatment as Usual: Children vs ImPACT at a Dose of 1 Hour/Week: Children; See protocol for full statistical analysis plan; Test type: Other; p = .04, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual: Children vs ImPACT at 4 Hours/Week: Children; See protocol for full statistical analysis plan; Test type: Other; p = .02, Regression, Linear

3. Primary Outcome: Early Intervention Parenting Self-Efficacy Scale (EIPSES)
Description: The EIPSES is a measure of parent self-efficacy. It is a 16-item self-report measure that examines parents beliefs about their ability to produce positive changes and promote optimal development in their child with a disability. Once items are summed, the total score ranges from 16-112, with higher scores indicating better self-efficacy and empowerment.
Time Frame: Baseline and 6 Month Follow Up (6 months)
Population: Participants in the arms/groups "Treatment as Usual: Early Interventionists", "ImPACT at a Dose of 1 Hour/Week: Early Interventionists", "ImPACT at 4 Hours/Week: Early Interventionists", "Treatment as Usual: Children", "ImPACT at a Dose of 1 Hour/Week: Children", "ImPACT at 4 Hours/Week: Children" are not included in the analysis as the measure's intent is to assess parent outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Caregivers
Number analyzed (Participants) | 12 | 17 | 17
score on a scale
  Baseline | 87.3 (9.7) | 84.8 (9.4) | 87.74 (6.14)
  Follow-Up | 87.5 (9.1) | 89.4 (12.2) | 89.95 (9.98)
Statistical Analysis 1: Comparison: Treatment as Usual: Caregivers vs ImPACT at a Dose of 1 Hour/Week: Caregivers; See protocol for full statistical analysis plan; Test type: Other; p = .78, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual: Caregivers vs ImPACT at 4 Hours/Week: Caregivers; See protocol for full statistical analysis plan; Test type: Other; p = .89, Regression, Linear

4. Primary Outcome: Parenting Interactions With Children: Checklist of Observations Linked to Outcomes (PICCOLO)
Description: Parent Responsiveness is measured using the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO™). PICCOLO is a checklist of 29 observable developmentally supportive parenting behaviors, with children ages 10-47 months, in four domains (affection, responsiveness, encouragement, and teaching).
  Each item is scored as 0, 1 or 2.
  0 = Behavior absent, not observed
  1. = Behavior barely there, sometimes
  2. = Behavior seen often
  Assessors add scores for each item to calculate a domain score and an overall domain score. Total scores can range from 0-58, with higher scores indicating more parent responsiveness to child behavior and actions.
Time Frame: Collected at Baseline and 6 Month Follow Up (time frame: 6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Caregivers
Number analyzed (Participants) | 12 | 17 | 17
total score on a scale
  Baseline | 35.5 (2.27) | 40.2 (2.10) | 38.0 (2.67)
  Follow-Up | 41.3 (2.24) | 36.8 (3.18) | 40.8 (2.57)
Statistical Analysis 1: Comparison: Treatment as Usual: Caregivers vs ImPACT at a Dose of 1 Hour/Week: Caregivers; See protocol for full statistical analysis plan; Test type: Other; p = .07, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual: Caregivers vs ImPACT at 4 Hours/Week: Caregivers; See protocol for full statistical analysis plan; Test type: Other; p = .88, Regression, Linear

5. Primary Outcome: Project ImPACT Intervention Fidelity Checklist
Description: Parent Treatment Adherence will be assessed through a videotaped parent-child interaction at home. Parent behavior will be scored for use of the intervention strategies using the Project ImPACT Intervention Fidelity Checklist. The scores range from 1 to 5, the higher the score representing the most adherence to the Project ImPACT intervention. The overall score is an average of scores from each item.
Time Frame: 6 months
Population: Treatment as Usual Children/Caregivers didn't receive the Project ImPACT intervention and not evaluated for their adherence to it. Participants in the arms/groups "Treatment as Usual: Early Interventionists", "ImPACT at a Dose of 1 Hour/Week: Early Interventionists", "ImPACT at 4 Hours/Week: Early Interventionists" are not included in the analysis as the measure's intent is to assess caregiver adherence to the intervention. A separate measure was used to evaluate interventionist's adherence.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Caregivers
Number analyzed (Participants) | 0 | 17 | 17
score on a scale |  | 2.8 (0.6) | 3.2 (0.7)

6. Primary Outcome: Project ImPACT Coaching Fidelity Checklist
Description: Clinician fidelity is measured using the Project ImPACT Coaching Fidelity Checklist. The checklist measures the providers' use of the core components to Project ImPACT. The form uses a 3-point score (scored from 0-2): 0, Not observed; 1, partially observed; and 2, observed. The final score is a summary percentage rating of overall fidelity with a range of 0-100%.
Time Frame: 3 Month Follow-Up (3 month time frame)
Population: Treatment as Usual providers did not implement Project ImPACT and were not evaluated using this fidelity measure. Participants in the arms/groups "Treatment as Usual: Families", "ImPACT at a Dose of 1 Hour/Week: Families", "ImPACT at 4 Hours/Week: Families" are not included in the analysis as the measure's intent is to assess the provider's adherence to the intervention. Parent adherence to the intervention was assessed with a separate measure.
Measure: Mean (Standard Deviation); unit: percentage of fidelity
Arm/Group | Treatment as Usual | ImPACT at a Dose of 1 Hour/Week | ImPACT at 4 Hours/Week
Number analyzed (Participants) | 0 | 6 | 6
percentage of fidelity |  | 55 (21) | 59 (24)

7. Primary Outcome: Vineland Adaptive Behavior Scales 3rd Edition-Socialization Domain
Description: The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.
  Because it is a norm-based instrument, the examinee's adaptive functioning is compared to that of others his or her age. The ABC score is based on scores for three specific adaptive behavior domains: Communication, Daily Living Skills, and Socialization.
  The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The standard score range for the Socialization domain is 20-140. Higher scores indicate better outcomes.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | ImPACT at a Dose of 1 Hour/Week | ImPACT at 4 Hours/Week
Number analyzed (Participants) | 12 | 17 | 17
score on a scale
  Baseline | 84.3 (12.2) | 76.4 (12.8) | 75.6 (15.0)
  Follow-Up | 78.7 (14.4) | 74.2 (19.0) | 70.1 (14.3)
Statistical Analysis 1: Comparison: Treatment as Usual vs ImPACT at a Dose of 1 Hour/Week; See protocol for full statistical analysis plan; Test type: Other; p = .26, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual vs ImPACT at 4 Hours/Week; See protocol for full statistical analysis plan; Test type: Other; p = .74, Regression, Linear

8. Secondary Outcome: Parent Empowerment and Coaching in Early Intervention (PEACE) Caregiver Coaching Fidelity Tool
Description: The PEACE Fidelity Tool measures a provider's caregiver coaching quality by evaluating the quality and use of evidence based caregiver coaching strategies during recorded EI session across 5 domains (collaboration, daily routines, demonstration, practice and feedback, and reflection).
  The tool consists of 25 items scored on a 5 point scale from 1-5. Domains and total scores are calculated by averaging items. Scores can range from 1-5, with higher scores indicating better coaching competency and quality.
Time Frame: 3 Month Follow Up (3 Months)
Population: Participants in the arms/groups "Treatment as Usual: Families", "ImPACT at a Dose of 1 Hour/Week: Families", "ImPACT at 4 Hours/Week: Families" are not included in the analysis as the measure's intent is to assess provider coaching fidelity.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual: Early Interventionists: The families keep receiving their treatment as usual
- ImPACT at a Dose of 1 Hour/Week: Early Interventionists: ImPACT at a dose of 1 hour/week over 6 months
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
- ImPACT at 4 Hours/Week: Early Interventionists: ImPACT at 4 hours/week over 6 months.
  Project ImPACT: Project ImPACT (Improving Parents As Communication Teachers) is an evidence-based parent-mediated intervention program based on best practices in early intervention. The program is designed for young children up to age six with social communication delays, including autism spectrum disorder. Project ImPACT focuses on social engagement, language, social imitation, and play. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI).
Arm/Group | Treatment as Usual: Early Interventionists | ImPACT at a Dose of 1 Hour/Week: Early Interventionists | ImPACT at 4 Hours/Week: Early Interventionists
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 2.8 (0.6) | 2.7 (0.4) | 2.6 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the course of 2 years for the study. Each participant's adverse event data was assessed during their study duration. For child/parent dyads, this was starting at Baseline and ending once they completed the 6 Month Followup assessment (6-7 month time period). For early interventionists, the adverse event period was starting at enrollment until all their enrolled child/parent dyads were finished with study procedures and their enrollment was complete (2 years)
Description: All unexpected adverse events were reported by study personnel to the DPH IRB and the IRB at Penn via standard adverse event reporting procedures. All adverse reactions were noted and discussed thoroughly with the PI, mentors, and IRB to determine proper reporting procedures on a case-by-case basis.
Arm/Group | Treatment as Usual: Children | Treatment as Usual: Early Interventionists | ImPACT at a Dose of 1 Hour/Week: Children | ImPACT at a Dose of 1 Hour/Week: Early Interventionists | ImPACT at 4 Hours/Week: Children | ImPACT at 4 Hours/Week: Early Interventionists | Treatment as Usual: Caregivers | ImPACT at a Dose of 1 Hour/Week: Caregivers | ImPACT at 4 Hours/Week: Caregivers
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/23 | 0/6 | 0/20 | 0/6 | 0/18 | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/23 | 0/6 | 0/20 | 0/6 | 0/18 | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/23 | 0/6 | 0/20 | 0/6 | 0/18 | 0/23 | 0/20

LIMITATIONS AND CAVEATS:
The study occurred during the height of the COVID-19 pandemic leading to additional stressors and burdens for participating providers and families.

High attrition in family participants occurred largely due to families dropping their services with their provider.

BOSCC video recordings were recorded in families' homes over Zoom, which introduced a high variability in quality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04729127/Prot_SAP_000.pdf